CLINICAL TRIAL: NCT04687020
Title: Long-term Use of Viltolarsen in Boys With Duchenne Muscular Dystrophy in Clinical Practice (VILT-502)
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: NS Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VILT-502
Record Dates: First submitted 2020-12-16; First posted 2020-12-29 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — viltolarsen

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Non-interventional (United States) / Low-interventional (Canada) : Viltolarsen (Other): Patients will receive viltolarsen (recommended dose 80mg/kg/week) during a treatment period up to 120 months.
  Interventions: Drug: Viltolarsen

INTERVENTIONS:
Drug: Viltolarsen — Received during weekly intravenous infusions

SUMMARY:
The VILT-502 study is Non-interventional Study(United States)/Low-intervention Clinical Trial (Canada) of Viltolarsen administered intravenously once weekly for 10 years to boys with DMD who complete the NS-065/NCNP-01-202 study.

DETAILED DESCRIPTION:
The VILT-502 study is an open-label, single-arm study to assess the long-term safety and effectiveness of viltolarsen, an exon skipping therapy for the treatment of DMD. Patients who complete the Phase II long-term extension study and meet the additional inclusion and exclusion criteria of the present protocol will be invited to enroll. Viltolarsen will be administered through weekly IV infusions, at the study site or at home.

The VILT-502 study will be conducted as a non-interventional study in the US, and as a low-intervention clinical trial in Canada where viltolarsen is not yet commercially available, owing to differences in the stage of regulatory approval in the two countries.

ELIGIBILITY:
Inclusion Criteria:

1. Patient, patient's parent or legal guardian have provided written informed consent/medical record release authorization prior to any extension study-specific procedures, and the patient has provided assent appropriate for his age and developmental status.
2. Patient completed the NS-065/NCNP-01-202 study and was judged by the investigator as appropriate to participate in the VILT-502 study.
3. Patient and parent or legal guardian are willing and able to comply with scheduled visits, study treatment administration plan, and study procedures.

Exclusion Criteria:

1. Patient has an allergy or hypersensitivity to the study drug or to any of its constituents.
2. Patient has severe behavioral or cognitive problems that preclude participation in the study, in the opinion of the investigator.
3. Patient has previous or ongoing medical condition, medical history, physical findings or laboratory abnormalities that could affect safety, make it unlikely that treatment and observation will be correctly completed or impair the assessment of study results, in the opinion of the investigator.
4. Patient had a treatment which was made for the purpose of dystrophin or its related protein induction after completing the NS-065/NCNP-01-202 study.
5. Patient took any other investigational drugs after completing the NS-065/NCNP-01-202 study.
6. Patient plans to participate in another clinical trial.
7. Patient was judged by the investigator and/or the Sponsor as not appropriate to participate in the study for reasons other than #1 - #6 above.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 9 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2032-09 (Estimated); Study Completion 2032-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment related Adverse Events as assessed by CTCAE v4.0 | baseline to up to 120 months of treatment
Change in Time to Stand (TTSTAND) | baseline to up to 120 months of treatment
Change in Time to Run/Walk 10 meters (TTRW) | baseline to up to 120 months of treatment
Change in Performance of Upper Limb (PUL) | baseline to up to 120 months of treatment
  The Performance of the Upper Limb (PUL) scale is a specifically designed for assessing upper limb function in ambulant and non-ambulant patients with DMD. It consists of 22 items subdivided into shoulder level (6 items), mid-level (9 items) and distal level (7 items) dimension. The item ranges from score 0 -no useful hand function -to score 6 full shoulder abduction.
Loss of Ambulation (LOA) | baseline to up to 120 months of treatment
  Loss of Ambulation (LOA) is defined by the inability to complete the Time to Run/Walk 10 meters (TTRW) in less than 30 seconds.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (4):
  - UC Davis, Sacramento, California
  - Lurie Children's Hospital, Chicago, Illinois
  - Duke University Medical Center, Durham, North Carolina
  - Children's Hospital of Richmond at VCU, Richmond, Virginia
- Alberta Children's Hospital, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Extension Study of NS-065/NCNP-01 in Boys With Duchenne Muscular Dystrophy (DMD) — https://clinicaltrials.gov/ct2/show/NCT03167255